CLINICAL TRIAL: NCT04451863
Title: Analgesic and Subjective Effects of Terpenes Administered Alone and in Combination With THC
Brief Title: Analgesic and Subjective Effects of Terpenes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-001519; R01AT010762-04 (NIH)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pain; Abuse, Drug
Keywords: Cannabis; Analgesia; Pain; THC; Terpenes
MeSH Terms: conditions — Pain; Substance-Related Disorders; Marijuana Abuse; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Placebo (Placebo Comparator): 0 mg THC, 0 mg myrcene, 0 mg BCP
  Interventions: Drug: Placebo
- Low strength THC (Active Comparator): 5 mg THC, 0 mg myrcene, 0 mg BCP
  Interventions: Drug: Low THC
- Higher strength THC (Active Comparator): 15 mg THC, 0 mg myrcene, 0 mg BCP
  Interventions: Drug: High THC
- Low strength myrcene (Active Comparator): 0 mg THC, 0.5 mg myrcene, 0 mg BCP
  Interventions: Drug: Low Myrcene
- High strength myrcene (Active Comparator): 0 mg THC, 12.0 mg myrcene, 0 mg BCP
  Interventions: Drug: High Myrcene
- Low strength BCP (Active Comparator): 0 mg THC, 0 mg myrcene, 0.5 mg BCP
  Interventions: Drug: Low Beta-Caryophyllene
- High strength BCP (Active Comparator): 15 mg THC, 0 mg myrcene, 7.5 mg BCP
  Interventions: Drug: High THC; Drug: High Beta-Caryophyllene
- Low THC + Low myrcene (Active Comparator): 5 mg THC, 0.5 mg myrcene, 0 mg BCP
  Interventions: Drug: Low THC; Drug: Low Myrcene
- Low THC + High myrcene (Active Comparator): 5 mg THC, 12.0 mg myrcene, 0 mg BCP
  Interventions: Drug: Low THC; Drug: High Myrcene
- High THC + Low myrcerne (Active Comparator): 15 mg THC, 0.5 mg myrcene, 0 mg BCP
  Interventions: Drug: High THC; Drug: Low Myrcene
- High THC + High myrcene (Active Comparator): 15 mg THC, 12.0 mg myrcene, 0 mg BCP
  Interventions: Drug: High THC; Drug: High Myrcene
- Low THC + Low BCP (Active Comparator): 5 mg THC, 0 mg myrcene, 0.5 mg BCP
  Interventions: Drug: Low THC; Drug: Low Beta-Caryophyllene
- Low THC + High BCP (Active Comparator): 5 mg THC, 0 mg myrcene, 7.5 mg BCP
  Interventions: Drug: Low THC; Drug: High Beta-Caryophyllene
- High THC + Low BCP (Active Comparator): 15 mg THC, 0 mg myrcene, 0.5 mg BCP
  Interventions: Drug: High THC; Drug: Low Beta-Caryophyllene
- High THC + High BCP (Active Comparator): 15 mg THC, 0 mg myrcene, 7.5 mg BCP
  Interventions: Drug: High THC; Drug: High Beta-Caryophyllene

INTERVENTIONS:
Drug: Low THC — Vaporized THC (5 mg)
  Arms: Low THC + High BCP; Low THC + High myrcene; Low THC + Low BCP; Low THC + Low myrcene; Low strength THC
Drug: High THC — Vaporized THC (15 mg)
  Arms: High THC + High BCP; High THC + High myrcene; High THC + Low BCP; High THC + Low myrcerne; High strength BCP; Higher strength THC
Drug: Low Myrcene — Vaporized Myrcene (0.5 mg)
  Arms: High THC + Low myrcerne; Low THC + Low myrcene; Low strength myrcene
Drug: High Myrcene — Vaporized Myrcene (12.0 mg)
  Arms: High THC + High myrcene; High strength myrcene; Low THC + High myrcene
Drug: Low Beta-Caryophyllene — Vaporized Beta-Caryophyllene (0.5 mg)
  Arms: High THC + Low BCP; Low THC + Low BCP; Low strength BCP
Drug: High Beta-Caryophyllene — Vaporized Beta-Caryophyllene (7.5 mg)
  Arms: High THC + High BCP; High strength BCP; Low THC + High BCP
Drug: Placebo — Vaporized Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to assess the analgesic and subjective effects of terpenes administered alone and in combination of THC.

DETAILED DESCRIPTION:
The overall aim of this placebo-controlled study is to examine dose-dependent analgesia, intoxication, abuse liability, and pharmacokinetics of ecologically relevant doses of vaporized myrcene and beta-caryophyllene administered alone or with vaporized THC.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 21-55 years
* Report non-medical use of cannabis 1-7 days per week over the 1 month prior to screening
* Not currently seeking treatment for cannabis use
* Urine test positive for recent cannabis use
* Have a Body Mass Index from 18.5 - 34kg/m2.
* Able to perform all study procedures
* Must be using a contraceptive method (hormonal or barrier methods)

Exclusion Criteria:

* Meeting DSM-V criteria for any substance use disorder other than nicotine, caffeine, or mild CUD
* Report using other illicit drugs in the prior 4 weeks
* • If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process not within the normal range and / or reveal any significant illness (e.g., hypertension) as judged by the study physician and to put the participant at greater risk of experiencing adverse events due to completion of study procedures.
* Current licit use of cannabis primarily for medical purposes, prescription analgesics, or any medications that may affect study outcomes
* Current pain
* Pregnancy is exclusionary due to the possible effects of the study medication on fetal development.
* History of an allergic reaction or adverse reaction to cannabis is exclusionary.
* History of respiratory illness or current respiratory illness
* History of seizure disorder or current seizure disorder
* Insensitivity to the cold water stimulus of the Cold Pressor Test
* Currently enrolled in another research protocol
* Current major Axis 1 disorders (mood, anxiety, or psychotic disorder)
* Not using a contraceptive method (hormonal or barrier methods)
* The evaluating physician reviews all medical assessments along with medical history. Any disorders that might make cannabis administration hazardous are exclusionary.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Analgesia as measured using the Cold Pressor Test | 7 hours
  Pain threshold and pain tolerance assessed using the Cold Pressor Test
Subject-rated drug effects of abuse liability | 7 hours
  Subject ratings of "Good Drug Effect" as measured using a visual analog scale (1-100 mm)

SECONDARY OUTCOMES:
Subject-rated drug effects of intoxication | 7 hours
  Subject ratings of "High" as measured using a visual analog scale (1-100 mm)
Subjective ratings of pain | 7 hours
  Subject ratings of Painfulness and Bothersomeness of the Cold Pressor Test

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No